CLINICAL TRIAL: NCT05542056
Title: Urinary Prostaglandin as a Potential Predictive Marker for Thiazide-induced Hyponatremia: a Prospective Cohort Study (The PROPHECY Study)
Brief Title: Urinary Prostaglandin as a Potential Predictive Marker for Thiazide-induced Hyponatremia
Acronym: PROPHECY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01241; kt21ChristCrain3
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Thiazide-induced Hyponatremia (TIH)
Keywords: Thiazide; Thiazide-like diuretics; Hyponatremia; Prostaglandin E2 (PGE2); Urinary PGE2 concentration; Plasma sodium level; Urinary prostaglandins
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and Urine aliquots are stored for eventual future research aims.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with newly prescribed thiazide or thiazide-like diuretic: As the study population of this observational study shall be as representative as possible all patients with a new thiazide or thiazide-like diuretic regardless of the indication, co-morbidities and co-medication can be included.
  Interventions: Other: Data and biosample collection

INTERVENTIONS:
Other: Data and biosample collection — Collection of spot urine, blood sampling, vital parameters, body weight, medical history, patient questionnaires, drinking protocol, drug diary at at Visit 1 (before thiazide initiation), at Optional 2 hours-challenge, at Visit 2 (4 weeks after thiazide initiation), at Visit 2.1 (4 weeks after dose change), at Visit 3 (3-months after thiazide initiation)

SUMMARY:
Thiazides and thiazide-like diuretics are one of the five major classes of antihypertensive drugs. This study is to investigate whether urinary PGE2 concentration at baseline (prior to thiazide initiation) is associated with the development of TIH within the first four weeks of treatment.

DETAILED DESCRIPTION:
Thiazides and thiazide-like diuretics are one of the five major classes of antihypertensive drugs. They act by inhibiting the apical Na+-Cl- -cotransporter in the distal convoluted tubules of the kidneys. Thiazides and thiazide-like diuretics often cause adverse effects, importantly a drop in plasma sodium levels that is called thiazide-induced hyponatremia (TIH). Data suggest a crucial role of urinary PGE2 in water reabsorption. Since urinary PGE2 concentrations were higher in patients with TIH, quantification of urinary PGE2 prior and after thiazide initiation might allow identification of patients at risk for TIH, presenting PGE2 as a potential novel predictive marker for the development of TIH.

This study is to investigate whether urinary PGE2 concentration at baseline (prior to thiazide initiation) is associated with the development of TIH within the first four weeks of treatment. Hospitalized and ambulatory patients in whom a thiazide or thiazide-like diuretic will be newly prescribed are screened for inclusion.

The study procedure contains the screening and inclusion, visit 1 before thiazide initiation, visit 2 4 weeks (+/-7days) after thiazide initiation and a 3-months follow-up (visit 3). An additional visit (visit 2.1) will only be added in case of a dose change of the thiazide or thiazide-like diuretic (4 weeks +/- 7 days after the dose change). The 2 hours- challenge is optional if the patient agrees to additional testing.

ELIGIBILITY:
Inclusion Criteria:

* Newly prescribed thiazide or thiazide-like diuretic
* ≥ 18 years of age
* Informed Consent as documented by signature

Exclusion Criteria:

* Intake of thiazide or thiazide-like diuretic in the preceding month
* Hyponatremia (plasma sodium <135 mmol/L) at baseline
* Acute infectious / inflammatory disease (CRP ≥ 20 mg/L [1, 11])
* Symptomatic urinary tract infection
* Chronic treatment with NSAID and / or NSAID intake 48 hours prior to urine sampling at visit 1 and 2 (intake of acetylsalicylic acid will be no exclusion criteria)
* End of life care, no informed consent or inability to follow the procedures of the study, e.g., due to language barriers, psychological disorders, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized and ambulatory patients in whom a thiazide or thiazide-like diuretic will be newly prescribed. Screening will take place at the University Hospital Basel and Kantonsspital Baselland, primarily at the Endocrine Outpatient Clinic and the Hypertension Clinic of the Medical Outpatient Clinic or Nephrology Department and is based on the patients' charts as well as consultation with the treating physician.
Sampling Method: Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of hyponatremia (plasma sodium <135 mmol/L) | Within the first four weeks of treatment (at visit 2)
  Occurrence of hyponatremia (plasma sodium <135 mmol/L)

SECONDARY OUTCOMES:
Change in urinary Prostaglandin- concentration | Between baseline, visit 2 (and visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in urinary Prostaglandin E2 (PGE2) and metabolite (PGE2M)- concentration
Change in the expression of proteins involved in sodium and water transport | Between baseline, visit 2 (and visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in the expression of proteins involved in sodium and water transport (AQP2, Prostaglandin transporter (PGT) and NCC) in urinary extracellular vesicles in spot urine (second morning urine)
Change in systolic and diastolic blood pressure | Between baseline, visit 2 (visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in systolic and diastolic blood pressure
Change in heart rate | Between baseline, visit 2 (visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in heart rate
Change in body weight | Between baseline, visit 2 (visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in body weight
Change in daily fluid intake | Between baseline, visit 2 (visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in daily fluid intake
Change in Bioelectrical impedance analysis (BIA) | Between baseline, visit 2 (visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in Bioelectrical impedance analysis (BIA)
Change in plasma sodium | Between baseline and visit 2 (and visit 2.1 if applicable), approximately 4 weeks
  Change in plasma sodium
Change in urine sodium | Between baseline and visit 2 (and visit 2.1 if applicable), approximately 4 weeks
  Change in urine sodium
Change in potassium | Between baseline and visit 2 (and visit 2.1 if applicable), approximately 4 weeks
  Change in potassium
Change in chloride | Between baseline and visit 2 (and visit 2.1 if applicable), approximately 4 weeks
  Change in chloride
Change in creatinine | Between baseline and visit 2 (and visit 2.1 if applicable), approximately 4 weeks
  Change in creatinine
Change in urea | Between baseline and visit 2 (and visit 2.1 if applicable), approximately 4 weeks
  Change in urea
Change in uric acid | Between baseline and visit 2 (and visit 2.1 if applicable), approximately 4 weeks
  Change in uric acid
Change in general well-being | Between baseline, visit 2 (visit 2.1 if applicable) and visit 3, approximately 3 months
  Change in general well-being rated on a visual analogue scale reaching from 0 to 10
Incidence of hyponatremia | Between baseline and visit 3, approximately 3 months
  Incidence of hyponatremia
Incidence of falls | Between baseline and visit 3, approximately 3 months
  Incidence of falls
Incidence of fractures | Between baseline and visit 3, approximately 3 months
  Incidence of fractures
Incidence of hospitalization due to any cause | Between baseline and visit 3, approximately 3 months
  Incidence of hospitalization due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — University Hospital Basel, Endocrinology, Diabetes and Metabolism
Locations (3):
- Hospital Universitario de Móstoles, Móstoles, Spain
- Switzerland (2):
  - University Hospital Basel, Endocrinology, Diabetes and Metabolism, Basel
  - Kantonsspital Baselland, Liestal